CLINICAL TRIAL: NCT04568018
Title: Open-label Trial to Assess the Efficacy and Safety of Inhalation Use of the Approved Drug Surfactant-BL (Biosurf LLC, Russia) as a Part of Complex Therapy of Acute Respiratory Distress Syndrome (ARDS) in Patients With SARS-CoV-2 Coronavirus Infection (COVID-19)
Brief Title: Surfactant-BL in Adult Acute Respiratory Distress Syndrome Due to COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Biosurf LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: Sur/ARDS-2020
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: ARDS Due to COVID-19
Keywords: Surfactant; ARDS; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Surface-Active Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1 cohort: Patients with mild ARDS, who are on spontaneous breathing.
  Patients who receive surfactant-BL through a mesh-nebulizer combined with the standard COVID-19 therapy, oxygen therapy according to the following scheme: inhalation of surfactant emulsion at 150 mg every 12 hours on the 1st, 2nd, 3rd, 4th and 5th days of the treatment period, inclusive.
  Interventions: Drug: Surfactant
- 2 cohort: Patients with moderate ARDS, who are on spontaneous breathing.
  Patients who receive surfactant-BL through a mesh-nebulizer combined with the standard COVID-19 therapy, oxygen therapy according to the following scheme: inhalation of surfactant emulsion at 150 mg every 12 hours on the 1st, 2nd, 3rd, 4th and 5th days of the treatment period, inclusive.
  Interventions: Drug: Surfactant
- 3 cohort: Patients with mild ARDS, receiving NIV and high-flow oxygen therapy.
  Patients who receive surfactant-BL through a mesh-nebulizer combined with the standard COVID-19 therapy, oxygen therapy, NIV and high-flow oxygen therapy according to the following scheme: inhalation of surfactant emulsion at 150 mg every 12 hours on the 1st, 2nd, 3rd, 4th and 5th days of the treatment period, inclusive.
  Interventions: Drug: Surfactant
- 4 cohort: Patients with moderate ARDS, receiving NIV and high-flow oxygen therapy.
  Patients who receive surfactant-BL through a mesh-nebulizer combined with the standard COVID-19 therapy, oxygen therapy, NIV and high-flow oxygen therapy according to the following scheme: inhalation of surfactant emulsion at 150 mg every 12 hours on the 1st, 2nd, 3rd, 4th and 5th days of the treatment period, inclusive.
  Interventions: Drug: Surfactant

INTERVENTIONS:
Drug: Surfactant — Inhalation of surfactant emulsion at 150 mg
  Other Names: Surfactant-BL

SUMMARY:
The purpose of this study is to prove the efficacy and safety Surfactant-BL, administered by inhalation in adult hospitalized patients with ARDS due to COVID-19.

DETAILED DESCRIPTION:
The efficacy and safety of Surfactant-BL will be evaluated in terms of mean duration of oxygen therapy (days) after hospitalization, in adult patients with ARDS due to SARS-COV-19 infection.

Adult patients with COVID-19 induced respiratory failure will be receive either standard treatment or standard treatment plus Surfactant-BL.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent for participation in the study.
2. Male of female ≥18 and ≤ 75 years of age.
3. Body-mass index (BMI) ≤ 40 kg/m2.
4. Probable (the presence of a characteristic clinical findings of COVID-19 in combination with characteristic changes in the lungs according to computer tomography (CT) data) or confirmed (according to the results of laboratory tests for the presence of SARS-CoV-2 RNA using nucleic acid amplification methods) diagnosis of COVID-19.
5. ARDS diagnosed within 24 hours prior to screening and confirmed at screening according to the following criteria (adapted Berlin criteria):

   * bilateral darkening of the pulmonary fields (infiltration, pulmonary edema) on the chest CT, which cannot be fully explained by pleural effusion, lung tissue atelectasis, tumor or other neoplasms;
   * nature of pulmonary infiltrates: respiratory failure not associated with heart failure or fluid overload;
   * oxygenation index (РаО2/FiO2 ratio): 150 mm hg < РаО2/FiO2 ≤ 300 mm hg at the positive end-expiratory pressure (PEEP) or the continuous positive air pressure (CPAP) ≥ 5 cm H2O.
6. Oxygen saturation of the blood according to pulseoximetry (SpO2) ≤ 93 % in ambient air.
7. No indications for immediate tracheal intubation and artificial lung ventilation (ALV).
8. Negative pregnancy test result (applicable to female patients with preserved breeding potential).

Exclusion Criteria:

1. ARDS due to the other viral infections.
2. Non-pulmonary ARDS.
3. Comorbidities continuing at the time of the screening or a history of comorbidities that increase the risk of patient transfer to ALV or may be fatal within 3 months, including but not limited to the following:

   * Any autoimmune diseases.
   * Resistant hypertension.
   * A history of stable ischemic heart disease, chronic heart failure (NYHA class III / IV) or unstable angina.
   * Congenital / acquired QT interval prolongation and / or history of the risk factors for QT interval prolongation.
   * Tuberculosis.
   * Suspected active uncontrolled bacterial, fungal, viral, or other infections (other than COVID-19).
   * Chronic kidney disease stage 4 or the need for hemodialysis / peritoneal dialysis.
   * Multiple organ dysfunction syndrome.
   * Cancer.
4. Patients with HIV infection, viral hepatitis B and C.
5. History of organ transplantation.
6. History of conditions requiring ALV.
7. Idiosyncrasy of study drug components.
8. Pregnancy, lactation.
9. Participation in any interventional clinical trial of any drug product at the time of the screening.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with ARDS due to SARS-COV-19 infection
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Mean duration of oxygen therapy (days) in the treatment group and in the control group. | within 5 days after the start of treatment

SECONDARY OUTCOMES:
The proportion of patients who required ALV within 5 days after the start of treatment. | within 5 days after the start of treatment
Change from baseline in PaO2/FiO2 ratio dynamics within 5 days after the start of treatment. | within 5 days after the start of treatment
Change from baseline in SpO2 dynamics within 5 days after the start of treatment. | within 5 days after the start of treatment
Proportion of patients who achieved an oxygenation index (PaO2/FiO2) of > 300 mm hg. | within 5 days after the start of treatment
Proportion of patients dead of any reason within 30 days after the start of treatment. | within 30 days after the start of treatment
Time to patient transfer to mechanically ventilated. | within 30 days after the start of treatment
Change from the baseline in the severity assessment of the patient's condition according to the NEWS-II scale within 5 days after the start of treatment. | within 5 days after the start of treatment
Change from baseline in leukocytes within 5 days after the start of treatment. | within 5 days after the start of treatment
Change from baseline in lymphocytes within 5 days after the start of treatment. | within 5 days after the start of treatment
Change from baseline in CRP within 5 days after the start of treatment. | within 5 days after the start of treatment
Change from baseline in ferritin within 5 days after the start of treatment. | within 5 days after the start of treatment
Change from baseline in D-dimer within 5 days after the start of treatment. | within 5 days after the start of treatment

OTHER OUTCOMES:
Rate of early terminations due to AE/SAE. | within 30 days after the start of treatment
Proportion of patients with AEs / SAEs with highly-reliable causal relationship (certain, probable or possible) with the current WHO therapy according to the researcher's opinion. | within 30 days after the start of treatment
Proportion of patients in each group with grade 3-4 AEs (CTCAE c 4.0 and higher) with highly-reliable causal relationship (certain, probable or possible) with the current WHO therapy according to the researcher's opinion. | within 30 days after the start of treatment
Proportion of deaths in each group. | within 30 days after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Avdeev, D.M.S., Principal Investigator — FSAEI of Higher Education I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- FSAEI of Higher Education I.M. Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided